CLINICAL TRIAL: NCT00004245
Title: A Phase I Study of Salicylate for Adult Patients With Advanced Myelodysplastic Disorders or Acute Myelogenous Leukemia
Brief Title: Sodium Salicylate in Treating Patients With Advanced Myelodysplastic Syndrome, Acute Myelogenous Leukemia, or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 99-057; P30CA008748 (NIH); MSKCC-99057; NCI-G99-1661
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; untreated adult acute myeloid leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Congenital Abnormalities | interventions — Sodium Salicylate

INTERVENTIONS:
Drug: sodium salicylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of sodium salicylate in treating patients who have advanced myelodysplastic syndrome , acute myelogenous leukemia or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the safety, toxicity, and pharmacokinetics of sodium salicylate in patients with advanced myelodysplastic syndrome; newly diagnosed, relapsed, or refractory acute myelogenous leukemia; or relapsed or refractory chronic lymphocytic leukemia.
* Define biologic characteristics that influence the likelihood of a clinical response to this drug in this patient population.

OUTLINE: Patients receive oral sodium salicylate twice a day. Intrapatient dose escalation or de-escalation is permitted. Treatment continues for up to 6 weeks in the absence of unacceptable toxicity or disease progression. Responding patients may continue to receive sodium salicylate beyond the 6-week period.

Patients with acute myelogenous leukemia are followed until the end of therapy. Patients with myelodysplastic syndrome are followed until death or progression to leukemia.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Relapsed or refractory acute myelogenous leukemia OR
* Elderly patients with newly diagnosed acute myelogenous leukemia not eligible for standard therapy OR
* "High-risk" myelodysplastic syndrome, including:

  * Refractory anemia with excess blasts
  * Refractory anemia with excess blasts in transformation
  * Chronic myelomonocytic leukemia OR
* Relapsed or refractory chronic lymphocytic leukemia
* Not eligible for transplant protocols at MSKCC or refuses transplant
* Not eligible for a higher priority protocol (e.g., bone marrow transplantation)

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 25,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* Transaminase levels less than 3 times upper limit of normal
* PT no greater than 14 seconds
* PTT no greater than 34.6 seconds

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Other:

* Not pregnant or nursing
* No history of abnormal bleeding or unexplained bleeding disorders
* No history of peptic ulcer disease
* No salicylate allergy
* No other concurrent active malignancy
* No other concurrent illness that would preclude study assessment to a significant degree

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Klimek, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Klimek VM, Dolezal EK, Smith L, Soff G, Nimer SD. Phase I trial of sodium salicylate in patients with myelodysplastic syndromes and acute myelogenous leukemia. Leuk Res. 2012 May;36(5):570-4. doi: 10.1016/j.leukres.2011.10.023. Epub 2011 Dec 9. PMID 22154022